CLINICAL TRIAL: NCT03401294
Title: Conversion From Unresectable To Resectable Liver Metastases In Patients With Liver-Only Metastatic Colorectal Cancer Treated With FOLFOXIRI Plus Bevacizumab. The Conversion Trial.
Brief Title: Conversion From Unresectable To Resectable Metastatic Colorectal Cancer.
Acronym: CONVERSION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Shahid Ahmed, Professor of Medicine, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99268
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Conversion therapy; Liver Metastasectomy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): FOLFOXIRI and Bevacizumab
  Interventions: Drug: FOLFOXIRI and Bevacizumab

INTERVENTIONS:
Drug: FOLFOXIRI and Bevacizumab — Every 2 week for a total of 12 cycles
  Other Names: 5FU, leucovorin, oxaliplatin, irinotecan and bevacizumab

SUMMARY:
Most patients with mCRC are treated with palliative chemotherapy and only a small number of patients with limited metastatic disease achieve long-term remission following metastasectomy. There is a growing need for more effective treatment in patients with liver-only mCRC to improve the rate of curative resection without compromising QOL.The current study is informed by our patient's needs. It aims to evaluate the rate of conversion therapy in patients with unresectable liver-only mCRC using the combination of FOLFOXIRI and bevacizumab and to assess the association between an early FDG-PT/CT response and other clinical and pathological biomarkers and hepatic metastasectomy.

DETAILED DESCRIPTION:
Colorectal cancer is the second leading cause of cancer-related death in North America. Patients with metastatic colorectal cancer generally have limited life expectancy, however, a small number of patients with liver-only metastases could potentially be cured following surgical resection of metastases. Patients and their family strongly feel that there is an unmet need for a more effective treatment in metastatic colorectal cancer to improve disease response rate and thereby curative surgery. Recent evidence suggest that a triplet chemotherapy regimen, FOLFOXIRI plus bevacizumab has been associated with higher response rates. The CONVERSION trial will evaluate the rate of conversion from unresectable to resectable liver metastases in patients with liver-only metastatic colorectal cancer treated with FOLFOXIRI-bevacizumab. Furthermore, this study will assess disease control rate, survival, quality of life and association between various biomarkers including an early FDG-PET/CT response and curative surgery. Thirty-two eligible patients will be recruited at the two major cancer centers in Saskatchewan. Patients will receive FOLFOXIRI-bevacizumab every two weeks for a total of 12 cycles and will undergo periodic imaging studies. The resectability of liver metastases will be assessed by a multidisciplinary team comprised of surgeons, radiologists, and oncologists. This study will be helpful to establish a standard chemotherapy regimen for patients with liver-only metastatic colorectal cancer and to determine the role of FDG-PET/CT scan and other biomarkers in predicting curative surgery. Complete resection of metastases will allow such patients to discontinue chemotherapy and live a normal life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged between 18 and 70 years with histologically proven adenocarcinoma or poorly differentiated carcinoma of the colon and rectum with unresectable liver-only metastases and no extra-hepatic disease.
* World Health Organization (WHO) performance status of 0-1.
* No previous chemotherapy for advanced disease.
* Adequate functioning of the bone marrow, liver, and kidneys.

Exclusion Criteria:

* Breastfeeding or pregnancy.
* An active second primary cancer with the exception of squamous cell carcinoma of the skin or an in situ cancer.
* Severe or uncompensated concomitant medical conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of liver metastasectomy | Up to 3 years from the date of enrolment into the study
  Conversion From Unresectable To Resectable Liver Metastases

SECONDARY OUTCOMES:
Response rate | Up to 12 weeks of last cycle of FOLFOXIRI from the date of enrolment till the date of maximum response
  Based on RECIST criteria
30 days rates of Grade III and IV toxicity | Up to 30 days of last cycle of FOLFOXIRI from the date of enrolment till the date of toxicity
  As per National Cancer Institute Common Toxicity Criteria
The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) | up to 3 years from the date of enrolment or till the progression of the disease
  Quality of life questionnaire related to cancer and its treatment
The European Organization for Research and Treatment of Cancer (EORTC) Colorectal Cancer Module (QLQ-CR29) | up to 3 years from the date of enrolment or till the progression of the disease
  Quality of life questionnaire specifically related to colorectal cancer
The European Organization for Research and Treatment of Cancer (EORTC) Colorectal Liver Metastases Module (LMC21) | up to 3 years from the date of enrolment or till the progression of the disease
  Quality of life questionnaire specifically related to liver metastases
Early-PET scan response | From the date of enrolment till 8 weeks after four cycles of FOLOXIRI and bevacizumab
  change in FDG-uptake between baseline and after 4 cycles of chemotherapy and it correlation with rate of metastasectomy
Progression-free survival | up to 5 years from the time of enrolment till disease progression or last follow up visit
  progression following FOLOXIRI and bevacizumab
Overall survival | up to 5 years from the time of enrolment till mortality or last follow up visit
  all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Ahmed, MD, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Allan Balir Cancer Center, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No